CLINICAL TRIAL: NCT05399381
Title: Precision Transcranial Electric Stimulation for the Therapy of Cognitive Impairment
Brief Title: Traveling-wave Transcranial Electric Stimulation
Acronym: TravelingTES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00002876; 30064 (Other Grant/Funding Number: Brain & Behavior Research Foundation)
Record Dates: First submitted 2022-04-06; First posted 2022-06-01 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Working Memory
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Frontoparietal Slow Theta Stimulation (Experimental): Participants will receive multi-electrode transcranial alternating current stimulation over the prefrontal and parietal brain regions that induces frontal-to-parietal traveling wave at the frequency of 4 Hz with the intensity of up to 2 mA and duration up to 20 min.
  Interventions: Device: Transcranial alternating current stimulation (tACS)
- Frontoparietal Fast Theta Stimulation (Experimental): Participants will receive multi-electrode transcranial alternating current stimulation over the prefrontal and parietal brain regions that induces frontal-to-parietal traveling wave at the frequency of 7 Hz with the intensity of up to 2 mA and duration up to 20 min.
  Interventions: Device: Transcranial alternating current stimulation (tACS)
- Parietofrontal Slow Theta Stimulation (Experimental): Participants will receive multi-electrode transcranial alternating current stimulation over the prefrontal and parietal brain regions that induces parietal-to-frontal traveling wave at the frequency of 4 Hz with the intensity of up to 2 mA and duration up to 20 min.
  Interventions: Device: Transcranial alternating current stimulation (tACS)
- Parietofrontal Fast Theta Stimulation (Experimental): Participants will receive multi-electrode transcranial alternating current stimulation over the prefrontal and parietal brain regions that induces parietal-to-frontal traveling wave at the frequency of 7 Hz with the intensity of up to 2 mA and duration up to 20 min.
  Interventions: Device: Transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: Transcranial alternating current stimulation (tACS) — Non-invasive, multi-electrode transcranial alternating current stimulation (tACS) over frontal and parietal brain areas.

SUMMARY:
This study will assess the impact of traveling wave transcranial alternating current stimulation (tACS) on working memory performance in adults.

DETAILED DESCRIPTION:
Transcranial alternating current stimulation (tACS) can non-invasively alter neuroelectric activity in the brain by applying weak time-varying electric currents via the scalp. Complex patterns of electric brain activity can take the form of traveling waves - spatially coherent brain rhythms that gradually propagate through the neocortex. Traveling waves are crucial for the temporal coordination of informational flow in the brain. Using the novel traveling-wave transcranial alternating current stimulation (tACS) approach, the investigators will explore the effects of frontal-to-parietal and parietal-to-frontal traveling waves on working memory performance and brain electrophysiology in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 45 years old.
2. Confident level of English language.

Exclusion Criteria:

1. History or evidence of chronic neurological or mental disorder.
2. Metal or electric implant in the head, neck, or chest area.
3. History of head injuries with loss of consciousness.
4. Any acute or chronic medical condition that requires ongoing pharmacological treatment.
5. Pregnancy or breast-feeding.
6. Alcohol or drug addiction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in working memory performance | Immediate effect during stimulation
  Changes in working memory performance (% of correct responses) as measured with the standardized N-back working memory task during active stimulation relative to pre-stimulation performance.

SECONDARY OUTCOMES:
Changes in reaction time | Immediate effect during stimulation
  Changes in reaction time (milliseconds) as measured using the standardized N-back working memory task during active stimulation relative to pre-stimulation performance.
Changes in electroencephalographic (EEG) connectivity | Five minutes post-stimulation
  Changes in electroencephalographic (EEG) connectivity in theta band (in normalized units) after transcranial electric stimulation relative to pre-stimulation periods.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Alekseichuk, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Full or partial access to the preprocessed data will be provided upon the request to the faculty / research staff of recognized research, medical, and educational institutions for educational and scientific purposes. The request should be sent via an institutional email and will be stored with the study materials. The request should include a short description of the scientific or educational aims.
Time Frame: Data will be shared only upon request after the study has ended (within 6 months).
Access Criteria: To receive access, the study investigators need to be contacted via an institutional e-mail including a short description of the scientific or educational aims.